CLINICAL TRIAL: NCT04678661
Title: My Dose Coach Titration and Maintenance in Patients With Type 2 Diabetes Mellitus on Basal Insulin
Brief Title: My Dose Coach Mobile App to Support Insulin Titration and Maintenance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues with app and prolonged recruitment
Sponsor: Linda Siminerio (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Linda Siminerio, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20040308
Record Dates: First submitted 2020-12-08; First posted 2020-12-22 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus Type 2 - Insulin-Treated
Keywords: Mobile application; Digital titration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- My Dose Coach (Insulin Dosing Support App) (Experimental): Phase 1 Titration: Patients receive insulin therapy education from diabetes educator (DE). Plus, DE trains patients to use My Dose Coach (MDC) for titration guidance according to an algorithm prepared by endocrinology provider (EP). Patients are asked to return for a 3-month (mo) follow-up clinic visit. Patients who successfully reach glycemic target are invited to Phase 2. Other patients are invited to continue titrating for another 3 months.
  Phase 2 Maintenance: At 3-mo clinic visit, an EP or DE trains patients the MDC Maintenance Module to support proper insulin dosing. Patients are asked to return for follow-up clinic visits at mo 6.
  Patients are surveyed (0, 3, 6 mo) to assess changes in behavioral and psychosocial factors that influence diabetes self-management and MDC acceptability.
  Interventions: Device: Smartphone application and web portal; Behavioral: Standard Insulin Therapy Education
- Usual Care Group (Active Comparator): A retrospective comparative group will be selected from eligible patients who previously were treated at the University of Pittsburgh Medical Center (UPMC) Diabetes Outpatient Clinics following standard insulin therapy education. Patients in the usual care group will be identified using data available in the electronic medical record system. Propensity score matching will be used to pair intervention and usual care participants during phase 1 of the study (baseline to 3 months).
  Interventions: Behavioral: Standard Insulin Therapy Education

INTERVENTIONS:
Device: Smartphone application and web portal — My Dose Coach is indicated for single patient use outside the clinic setting by a previously diagnosed Type 2 Diabetic who has been prescribed a once-daily long-acting basal insulin. MDC is intended as an aid to the patient to provide dose suggestions based upon the HCP's independent professional judgment. Before My Dose Coach can be used, the HCP configures the dose instructions for the specific patient and activates the application using the specific patient Instructions. The application uses the dose plan instructions provided by the patient's HCP to provide dose suggestions of once-daily long-acting basal insulin (i.e. basal insulin titration) that are based on the patient's Fasting Blood Glucose (FBG) as well as hypoglycemia occurrence.
  MDC includes a Maintenance Module designed to support patients in maintaining proper insulin dosingby enabling logging of administered doses of prescribed diabetes medications and BGM and providing dosing and measurement reminders.
  Other Names: My Dose Coach
  Arms: My Dose Coach (Insulin Dosing Support App)
Behavioral: Standard Insulin Therapy Education — Standard best practices for training patients to administer insulin therapy include 1) a thorough patient assessment prior to therapy initiation to address barriers, including evaluation for diminished cognitive capacity or other problem that may impair safe insulin self-administration, and assessment of health literacy and numeracy skills; 2) observation of a patient's injection practice, with re-education provided as needed; 3) use of appropriate language is necessary when teaching injection technique; 4) dose preparation, which includes inspecting the insulin dose for accuracy (following manufacturer instructions); and 5) review of signs, symptoms and treatment of hypoglycemia must be included as a critical component of the training.

SUMMARY:
The purpose of this research study is to evaluate an electronic application (app) designed to help people with type 2 diabetes (T2DM) adjust their insulin doses. The app is called My Dose Coach. This research study is being done in 2 phases. Specifically in Phase 1, the study is assessing the role of the My Dose Coach app in helping participants make insulin adjustments to get their blood glucoses to the target level that is planned for with the diabetes team, called the dosing or titration phase, when first starting insulin. In Phase 2, the study is assessing the role of the My Dose Coach app in helping participants keep blood glucoses in the target range, called the maintenance phase.

DETAILED DESCRIPTION:
Despite the increasing body of knowledge of diabetes treatment strategies, a majority of patients with T2DM are still in a persistent state of poor glycemic control and unable to meet target goals. Inertia surrounding insulin initiation and titration is a specific problem. Various approaches have been proposed to help overcome clinical inertia, including support of patient self-management, and education for both physicians and people with diabetes. Presently, paper-based guides are available in which clinicians/educators rely on to help their patients in determining and recording appropriate insulin doses. Unfortunately, this process often sets the stage for reluctance and fear of insulin initiation and delays titration with implications for long-term poor self-management and adherence. Therefore, Sanofi developed the My Dose Coach electronic app to assist with optimizing titration of basal insulins and supporting proper insulin maintenance. The primary objective of this two phase study is to demonstrate that patients who are trained on the My Dose Coach app to titrate insulin will have greater improvements in hemoglobin A1c and will be more likely to achieve glycemic control at three months as compared to usual care practice, and, for the intervention group only, those who do attain glycemic goals will be able to maintain glycemic control for an additional three months. The secondary objective of this study is to examine the feasibility of integrating digital solutions into clinical workflow and user acceptability of My Dose Coach.

ELIGIBILITY:
Inclusion Criteria:

Intervention Group

* Patient receiving care at a UPMC Diabetes Outpatient and/or Inpatient settings
* Adult male and female patients 18 to 75 years old
* HbA1c > 7.5%
* Recommended to start self titration of basal insulin
* Access to and able to use an iOS (Apple phone operating system) or Android enabled device and have reliable internet access
* Willing and able to use the MDC app
* Able to comprehend basic diabetes survival skills, signs and symptoms of hypoglycemia and treatment of BG

Usual Care Group

* Adult male and female patients 18 to 75 years old
* HbA1c > 7.5%
* Started on basal insulin in a UPMC Diabetes Outpatient facility within the past three years of study start
* Has blood glucose data available in electronic medical records (EMR) (At least two HbA1c measurements corresponding to baseline and a subsequent time point after insulin titration)

Exclusion Criteria:

* Pregnant or breastfeeding
* Patients unwilling to use MDC app

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Siminerio, RN, PhD, CDE, Principal Investigator — Professor
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A consent form used in enrolling participants will be posted.
Supporting Information: ICF
Time Frame: After the clinical trial is closed to recruitment, and no later than 60 days after the last study visit by any subject, as required by the protocol.
Access Criteria: ICF will be added to Clinicaltrials.gov record.

REFERENCES:
- [Result] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Result] Fisher L, Hessler DM, Polonsky WH, Mullan J. When is diabetes distress clinically meaningful?: establishing cut points for the Diabetes Distress Scale. Diabetes Care. 2012 Feb;35(2):259-64. doi: 10.2337/dc11-1572. Epub 2012 Jan 6. PMID 22228744
- [Result] Peyrot M, Xu Y, Rubin RR. Development and validation of the Diabetes Medication System Rating Questionnaire-Short Form. Diabet Med. 2014 Oct;31(10):1237-44. doi: 10.1111/dme.12453. Epub 2014 Apr 18. PMID 24673614

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified at participating community-based primary care practices, diabetes outpatient clinics and hospital inpatient units.
Pre-assignment Details: Usual care is a historical comparison group, therefore usual care participants were not considered to be enrolled into the study.
Groups:
- My Dose Coach (Insulin Dosing Support App): Phase 1 Titration: Patients received insulin therapy education from diabetes educator (DE) and were trained to use the My Dose Coach (MDC) app for titration guidance according to an algorithm prepared by endocrinology provider (EP). Patients were asked to return for a 3-month (mo) follow-up clinic visit. Patients who successfully reached glycemic target were invited to Phase 2. Those who did not reach glycemic target were invited to continue titrating with the app for another 3 mo.
  Phase 2 Maintenance: At 3-mo clinic visit, an EP or DE trained patients the MDC Maintenance Module to support proper insulin dosing for another 3 mo.
  Patients were surveyed (0, 3, 6 mo) to assess changes in behavioral and psychosocial factors that influence diabetes self-management and MDC acceptability.
- Usual Care Group: A retrospective comparative group was be selected from eligible patients who previously were treated at the University of Pittsburgh Medical Center (UPMC) Diabetes Outpatient Clinics following standard insulin therapy education. Patients in the usual care group were identified using data available in the electronic medical record system. Propensity score matching were used to pair intervention and usual care participants.
Period: Overall Study
Arm/Group | My Dose Coach (Insulin Dosing Support App) | Usual Care Group
Started | 60 | 33
Completed | 36 | 33
Not Completed | 24 | 0
Not completed — Study paused to address technical issues related to the app. Participants removed from study . | 17 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Population: Usual care participants were identified through retrospective chart review; they were not formally enrolled in the study.
Groups:
- Intervention: Phase 1 Titration: Patients received insulin therapy education from diabetes educator (DE) and were trained to use the My Dose Coach (MDC) app for titration guidance according to an algorithm prepared by endocrinology provider (EP). Patients were asked to return for a 3-month (mo) follow-up clinic visit. Patients who successfully reached glycemic target were invited to Phase 2. Those who did not reach glycemic target were invited to continue titrating with the app for another 3 mo.
  Phase 2 Maintenance: At 3-mo clinic visit, an EP or DE trained patients the MDC Maintenance Module to support proper insulin dosing for another 3 mo.
  Patients were surveyed (0, 3, 6 mo) to assess changes in behavioral and psychosocial factors that influence diabetes self-management and MDC acceptability.
- Usual Care: A retrospective comparative group was be selected from eligible patients who previously were treated at the University of Pittsburgh Medical Center (UPMC) Diabetes Outpatient Clinics following standard insulin therapy education. Patients in the usual care group were identified using data available in the electronic medical record system. Propensity score matching were used to pair intervention and usual care participants.
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 60 | 33 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 27 | 73
  >=65 years | 14 | 6 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 20 | 53
  Male | 27 | 13 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 55 | 33 | 88
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 52 | 31 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 33 | 93
Hemoglobin A1c [Mean (Standard Deviation); unit: % glycated hemoglobin] | 9.8 (1.7) | 9.7 (1.4) | 9.8 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycemic Control at 3 Months
Description: Average change in hemoglobin A1c from baseline to 3 months
Time Frame: Baseline to 3 months
Population: Using propensity score matching, 33 intervention participants were paired with 33 usual care participants to compare changes in hemoglobin A1c from baseline to 3 months.
Measure: Mean (Standard Deviation); unit: % glycated hemoglobin
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 33 | 33
% glycated hemoglobin | -2 (2.2) | -1.7 (1.9)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = .207, Regression, Linear — Propensity score matching was used to form pairs of intervention and control participants. Specifically, a greedy matching procedure with a matching caliper of 0.2 of the standard deviation of the logit of the propensity score was used; Model adjusted for covariates of age, race, baseline BMI, and baseline hemoglobin A1c

2. Secondary Outcome: Change From Baseline in Fasting Blood Glucose at 3 Months
Description: Change in fasting blood glucose from baseline to 3 months for the intervention group.
Time Frame: Baseline to 3 months
Population: Population includes all intervention participants who completed the study and had fasting blood glucose values at both baseline and 3 month timepoints. Fasting blood glucose values were not collected for the historic usual care group so they were not included for analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention
Number analyzed (Participants) | 31
mg/dL | -33.4 (68.2)
Statistical Analysis 1: Comparison: Intervention; Independent t-test; Test type: Other; p = .011, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose at 6 Months
Description: Change in fasting blood glucose from baseline to 6 months for the intervention group.
Time Frame: Baseline to 6 months
Population: Participants in the intervention group who completed the study and had fasting blood glucose values recorded at time points of comparison. Data were not collected for the historic usual care group so they were not included for analysis of this outcome.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Intervention
Number analyzed (Participants) | 25
mg/dl | -38.3 (79.8)
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = .024, t-test, 2 sided

4. Secondary Outcome: Change From 3 Months in Fasting Blood Glucose at 6 Months
Description: Chang in fasting blood glucose from month 3 to 6 for the intervention group.
Time Frame: Months 3 to 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention
Number analyzed (Participants) | 23
mg/dL | 5 (42.6)
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = .579, t-test, 2 sided

5. Secondary Outcome: Change From Baseline in Hemoglobin A1c at 6 Months
Description: Average change in hemoglobin A1c from baseline to 6 months for the intervention group.
Time Frame: Baseline to 6 months
Population: All participants in the intervention group with available hemoglobin A1 data at the specified time points were included. Data were not collected for the historic usual care group so they were not included for analysis of this outcome.
Measure: Mean (Standard Deviation); unit: % glycated hemoglobin
Arm/Group | Intervention
Number analyzed (Participants) | 34
% glycated hemoglobin | -2.3 (2.3)
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p < .001, t-test, 2 sided — Reported p-value was calculated

6. Secondary Outcome: Change From 3 Months in Hemoglobin A1c at 6 Months
Description: Average change in hemoglobin A1c from 3 months to 6 months for the intervention group.
Time Frame: Months 3 to 6
Population: All participants in the intervention group who had hemoglobin A1c values available at time points of comparison were included. Data were not collected for the historic usual care group so they were not included for analysis for this outcome.
Measure: Mean (Standard Deviation); unit: % glycated hemoglobin
Arm/Group | Intervention
Number analyzed (Participants) | 31
% glycated hemoglobin | -.16 (.8)
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = .269, t-test, 2 sided

7. Secondary Outcome: Proportion of Patients Who Achieve Glycemic Targets
Description: Achieving glycemic target defined as reduction in hemoglobin A1c <7% by 3 months after baseline
Time Frame: 3 months
Population: Intervention group includes those participants who completed the study and had 3 month hemoglobin A1c values. Usual care is a historical comparative group.
Measure: Number; unit: proportion of participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 32 | 33
proportion of participants | .31 | .3

8. Secondary Outcome: Proportion of Patients Who Maintain Glycemic Targets
Description: Maintaining glycemic target defined as maintaining a hemoglobin A1c <7% at 6 months for those who achieved this target at 3 months in the intervention group.
Time Frame: 6 months
Population: Participants in the intervention group who reached their target glycemic goal (hemoglobin A1c <7%) at 3 months and had hemoglobin A1c values available at 6 months. Data were not collected for the historic usual care group so they were not included for analysis for this outcome.
Measure: Number; unit: proportion of participants
Arm/Group | Intervention
Number analyzed (Participants) | 10
proportion of participants | 1

9. Secondary Outcome: Change From Baseline in Diabetes Distress at 3 Months
Description: Diabetes distress was evaluated with the 17-item Diabetes Distress Scale, which assesses four dimensions of distress - emotional, regimen, interpersonal and physician, and has shown a consistent pattern of relationships with HbA1c, diabetes self-efficacy, diet and physical activity in multiple samples of patients with T2DM. Individual items are scored from 1 to 6; total scores are the average of all individual item scores; higher scores indicate greater distress. Possible scores range from 1 to 6.
Time Frame: Baseline to 3 months
Population: All participants in the intervention group who completed the study. Data were not collected for the historic usual care group so they were not included for analysis for this outcome.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Intervention
Number analyzed (Participants) | 36
Score on scale | -.47 (.55)
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p < .001, t-test, 2 sided — Reported p-value was calculated

10. Secondary Outcome: Change From Baseline in Diabetes Distress at 6 Months
Description: as for outcome 9
Time Frame: Baseline to 6 months
Population: All intervention participants who completed the study. Data were not collected for the historic usual care group so they were not included for analysis for this outcome.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Intervention
Number analyzed (Participants) | 36
Score on scale | -.49 (.57)
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p < .001, t-test, 2 sided — Reported p-value was calculated

11. Secondary Outcome: Change From 3 Months in Diabetes Distress at 6 Months
Description: as for outcome 9
Time Frame: Month 3 to month 6
Population: All participants who completed the intervention. Data were not collected for the historic usual care group so they were not included for analysis for this outcome.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Intervention
Number analyzed (Participants) | 36
Score on scale | -.02 (.3)
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = .647, t-test, 2 sided

12. Secondary Outcome: Participant Acceptability of Insulin Dosing Support System for Insulin Titration
Description: Participants rated their acceptability of My Dose Coach using a study-specific survey. Individual items are scored from 1 to 5; total scores are the average of all individual item scores; . Possible score range 1 to 5. The higher the score, the better the rating or acceptability of the insulin dosing support system.
Time Frame: 3 months
Population: All participants in the intervention who completed the study.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Intervention
Number analyzed (Participants) | 36
Score on scale | 4.6 (.7)

13. Secondary Outcome: Participant Satisfaction With Insulin Treatment
Description: The Diabetes Medication Systems Rating Questionnaire-Short Form, was also be used to inform patient acceptability and satisfaction with insulin. This questionnaire includes 20 items to assess convenience, negative events, interference, self-monitoring of blood glucose burden, efficacy, social burden, psychological well-being, treatment satisfaction and treatment preference. All items are scored 0 to 100. Composite score is calculated as means of completed items. Possible score range is 0 to 100. The higher the score, the higher the level of satisfaction.
Time Frame: 6 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Intervention
Number analyzed (Participants) | 36
Score on scale | 82.6 (10.9)

14. Secondary Outcome: Number of Hypoglycemic Events
Description: Total number of hypoglycemic events where blood glucose <70mg/dl.
Time Frame: As reported across study period, up to 6 months
Population: All participants in the intervention who completed the study. Did not collect on historic control group.
Measure: Number; unit: Events
Arm/Group | Intervention
Number analyzed (Participants) | 36
Events | 15

15. Secondary Outcome: Number of Participants Who Experienced Severe Hypoglycemic Events.
Description: Severe hypoglycemic events were defined a hypoglycemic events that required assistance of another person to resuscitate because blood glucoses are too low to maintain consciousness.
Time Frame: As reported across study period, up to 6 months
Population: All participants in the intervention who completed the study. Did not collect on historic control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 36
Participants | 0

16. Other Pre Specified Outcome: Participant Use of My Dose Coach
Description: Patient use of My Dose Coach app was track through the app's data analytics software platform. High app use was defined as logging in app >3days per week.
Time Frame: As reported across study period, up to 6 months
Population: All intervention participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 36
Participants | 11

17. Other Pre Specified Outcome: Number of Technical Complaints
Description: Number of technical complaints made by participants about My Dose Coach app
Time Frame: As reported across study period, up to 6 months
Population: All participants enrolled in intervention.
Measure: Number; unit: Number of complaints
Arm/Group | Intervention
Number analyzed (Participants) | 60
Number of complaints | 20

18. Other Pre Specified Outcome: Frequency of Escalation of Care
Description: Frequency of endocrinology and other medical visits beyond protocol will be used to assess escalation of care
Time Frame: As reported across study period, up to 6 months
Population: All participants enrolled in the intervention. Data were not collected for the historic usual care group so they were not included for analysis for this outcome.
Measure: Number; unit: Number of visits
Arm/Group | Intervention
Number analyzed (Participants) | 60
Number of visits | 0

19. Other Pre Specified Outcome: Type of Technical Complaints
Description: Type of technical complaints made by participants about My Dose Coach app
Time Frame: As reported across study period, up to 6 months
Population: All participants enrolled in intervention
Measure: Number; unit: Type of complaints
Arm/Group | Intervention
Number analyzed (Participants) | 60
Type of complaints | 15

20. Other Pre Specified Outcome: Type of Escalation of Care
Description: Type of endocrinology and other medical visits beyond protocol were used to assess escalation of care
Time Frame: As reported across study period, up to 6 months
Population: All patients enrolled in the intervention. Did not collect on historic control group.
Measure: Number; unit: Type of escalation of care
Arm/Group | Intervention
Number analyzed (Participants) | 60
Type of escalation of care | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/60 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/33
Other Adverse Events (participants affected / at risk) | 15/60 | 0/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=60) | Usual Care (N=33)
Mild Hypoglycemic Event (Endocrine disorders) | 15 (15) | 0 (0) — Mild/asymptomatic hypoglycemia - blood glucose <70 mg/dl and no symptoms

LIMITATIONS AND CAVEATS:
The trial was implemented during the COVID-19 pandemic and there were restrictions and challenges with meeting enrollment goals. Early on in the study, a technical issue with the intervention app was discovered and required that the study be paused while the issue was addressed, further impacting enrollment goals. Also, the study design included a historic control group to make best use of available resources, which limited comparisons among study groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT04678661/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT04678661/ICF_001.pdf